CLINICAL TRIAL: NCT02921282
Title: Nicotine Reinforcement and Smoking-Cue Reactivity: Association With Genetic Polymorphisms
Status: Completed | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Bernard Le Foll, Scientist, Centre for Addiction and Mental Health
Other Study IDs: 134-2015
Record Dates: First submitted 2016-09-22; First posted 2016-10-03 (Estimated); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Cigarette Smoking Behavior
Keywords: genes; cues; reward; smoking
MeSH Terms: conditions — Cigarette Smoking; Smoking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Genotype dopamine: Genotyping will be conducted at the conclusion of the study
  Interventions: Genetic: Genotype dopamine; Genetic: Genotype cannabinoids
- Genotype cannabinoids: Genotyping will be conducted at the conclusion of the study
  Interventions: Genetic: Genotype dopamine; Genetic: Genotype cannabinoids

INTERVENTIONS:
Genetic: Genotype dopamine — Laboratory investigations of nicotine reinforcement
Genetic: Genotype cannabinoids — Laboratory investigations of nicotine reinforcement

SUMMARY:
In this study, potential associations between several genetic polymorphisms and nicotine dependence will be examined. The relative reinforcing efficacy of cigarettes using the forced-choice procedure will be assessed. In addition, reactivity to smoking cues using a reliable procedure will be conducted.

DETAILED DESCRIPTION:
It is known that cannabinoid and dopamine receptors can be important modulators of response to nicotine and its associated cues. In this study participants will be genotyped to determine whether there is a relationship between CB1 or D3 genes and the reinforcing properties of nicotine or the subjective effects of nicotine-associated cues. In one session, participants will chose between two different cigarettes, each with different properties. In another session, physiological responses and craving will be measured when presented with cues that remind participants of nicotine. At some point during the study, blood will be collected for genotyping and this will processed to study whether CB1 or D3 genotype influences these responses to nicotine or cues.

ELIGIBILITY:
Inclusion Criteria:

1. 19-64 year old males and females
2. smoking at least 10 cigarettes per day for at least 1 year
3. positive urinary cotinine
4. medically and psychologically healthy as determined by screening criteria

Exclusion Criteria:

1. definite plan to reduce or quit tobacco use during the course of the study
2. treatment for tobacco dependence in the past 3 months
3. use of nicotine replacement products, bupropion, or varenicline in the past 3 months
4. consumption of more than 15 alcoholic drinks per week during the past month
5. use of any illicit drug more than twice per week during the past month
6. current use of any medication that would interfere with the protocol in the opinion of PI
7. under the influence of a drug or alcohol at any session
8. pregnant, nursing, or become pregnant during the study

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Otherwise healthy smokers will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Number of puffs on a cigarette | 3 years
  Puffs taken from either a nicotinized or a denicotinized cigarette

SECONDARY OUTCOMES:
Craving in response to nicotine cues | 3 years
  Craving scores measured by questionnaires in response to either smoking-related or neutral cues
Physiological measures in response to cues | 3 years
  Physiological measures (eg., heart rate and/or blood pressure) in response to smoking-related or neutral cues

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD PhD, Principal Investigator — CAMH
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No